CLINICAL TRIAL: NCT06027489
Title: The Effect of Listening to Music and Drawing on the Coping With Dysmenorrhea of Nursing Students Experiencing Dysmenorrhea
Brief Title: Listening Music, Drawing on Coping With Dysmenorrhea Complaints of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Assist. Prof, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/SBB/0415
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Music; Drawing; Coping Behavior; Dysmenorrhea; Symptom, Depressive; Dysmenorrhea Symptom
Keywords: Music; Drawing; Nursing Students; Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea; Depression | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Nursing students with dysmenorrhea in the control group were informed that drawing and listening to music practices would be performed after the initial, second and third month evaluations of the study. In the meantime, it was stated that he should not make any interventions other than her routine applications. At baseline, second, and third month, participants will measure pain, menstrual symptoms, and perceived stress on the first day of the menstrual cycle using the VAS, MSS, and PSS, respectively.
- Music Group (Experimental): In the second and third months, participants listened to a song that lasted 29 minutes and 32 seconds for four days (three days before menstruation and the first day of menstruation). The song to be played was determined by examining the literature, the song was composed by researcher Juan Sebastian Martin-Saavedra and was named Occasio Adolore (Music Piece No. 5-559-355 and Phonogram No. 12-105-295) by the author copyright institution of Colombia. registered under. While the researcher is composing the song, it is to create a piece of music that will reduce the pain felt, activate positive emotions and relax the person. The composed song is available online within the scope of the published article (https://soundcloud.com/jss-martin/occasio-adolore) [21]. Written permission was obtained from Juan Sebastian Martin-Saavedra to use the composed song in the research. The access link of the composed song will be sent to the participants via social media (WhatsApp).
  Interventions: Behavioral: Music
- Drawing Group (Experimental): In the second and third months, the participants will be asked to paint for 29 minutes and 32 seconds (the duration of the intervention was determined in parallel with the music group in order not to create variability between the groups) for four days (three days before menstruation and the first day of menstruation). The type of paint to be used in the drawn picture (dry pen, crayon or watercolor) is left to the availability of the participants, and it will be stated that they prefer colors and drawings that will raise their emotions, focus their drawings and feed positive emotions in the picture to be drawn. After drawing pictures three days before the menstrual cycle and the first day of menstruation (for a total of four days), pain, menstrual symptoms, and perceived stress on the first day of menstruation will be measured using the VAS, MSS, and PSS, respectively.
  Interventions: Behavioral: Drawing Group

INTERVENTIONS:
Behavioral: Music — In the second and third months, participants listened to a song that lasted 29 minutes and 32 seconds for four days (three days before menstruation and the first day of menstruation). The song to be played was determined by examining the literature, the song was composed by researcher Juan Sebastian Martin-Saavedra and was named Occasio Adolore (Music Piece No. 5-559-355 and Phonogram No. 12-105-295) by the author copyright institution of Colombia. registered under. While the researcher is composing the song, it is to create a piece of music that will reduce the pain felt, activate positive emotions and relax the person. The composed song is available online within the scope of the published article (https://soundcloud.com/jss-martin/occasio-adolore).
  Arms: Music Group
Behavioral: Drawing Group — : In the second and third months, the participants will be asked to paint for 29 minutes and 32 seconds (the duration of the intervention was determined in parallel with the music group in order not to create variability between the groups) for four days (three days before menstruation and the first day of menstruation). The type of paint to be used in the drawn picture (dry pen, crayon or watercolor) is left to the availability of the participants, and it will be stated that they prefer colors and drawings that will raise their emotions, focus their drawings and feed positive emotions in the picture to be drawn.
  Arms: Drawing Group

SUMMARY:
Objectives: Investigating the effects of listening to music and drawing on nursing students with dysmenorrhea on dysmenorrhea complaints is a new and promising area of research. However, high-level evidence on whether listening to music and drawing has an effect on dysmenorrhea complaints is insufficient. The current study addresses this research question..

Design: A three-arm randomized controlled trial was conducted in 96 nursing students with dysmenorrhea.

DETAILED DESCRIPTION:
This three-armed randomized controlled study (RCT) will be conducted in July 2023 in Bartın University Faculty of Health Sciences Nursing Department students experiencing dysmenorrhea. Nursing students who experienced dysmenorrhea at the time of application were informed about the aims, setup and intervention of the study. and evaluated for suitability in a short, standardized interview. Nursing students experiencing dysmenorrhea who met our criteria were given a basic questionnaire along with a letter of information and an informed consent form. Nursing students with dysmenorrhea gave written informed consent for participation in the study were included. Evaluations in all three groups were made before randomization (ie baseline) and immediately after the intervention periods (2nd and 3rd month).

Randomization: The randomization list was made by another scientist who was not involved in the research process in order to preserve the random selection order and to prevent bias, and with this blinding applied, the group allocation was hidden. A computer randomization program was used to generate the randomization list for the intervention allocation sequence. Individuals who received a voluntary consent form and volunteered to participate in the research were randomly assigned to the experimental and control groups by using the blocking method. Following simple randomization procedures, participants were assigned to one of the three arms of the study in a 1:1:1 ratio according to a computer-generated randomization scheme via https://www.sealedenvelope.com/simple-randomiser/v1.

In this research, the allocation of participants to groups was made by scientists who were not involved in the research. Due to the nature of the research, the follow-up of the practices and the participants will not be provided during the data collection process, as the researcher does it.

Intervention:

Music Group: In the second and third months, participants listened to a song that lasted 29 minutes and 32 seconds for four days (three days before menstruation and the first day of menstruation). The song to be played was determined by examining the literature, the song was composed by researcher Juan Sebastian Martin-Saavedra and was named Occasio Adolore (Music Piece No. 5-559-355 and Phonogram No. 12-105-295) by the author copyright institution of Colombia. registered under. While the researcher is composing the song, it is to create a piece of music that will reduce the pain felt, activate positive emotions and relax the person. The composed song is available online within the scope of the published article (https://soundcloud.com/jss-martin/occasio-adolore). Written permission was obtained from Juan Sebastian Martin-Saavedra to use the composed song in the research. The access link of the composed song will be sent to the participants via social media (WhatsApp). After listening to music for three days before the menstrual cycle and on the first day of menstruation (for a total of four days), pain, menstrual symptoms and perceived stress on the first day of menstruation will be measured using VAS, MSS, and PSS, respectively.

Drawing Group: In the second and third months, the participants will be asked to paint for 29 minutes and 32 seconds (the duration of the intervention was determined in parallel with the music group in order not to create variability between the groups) for four days (three days before menstruation and the first day of menstruation). The type of paint to be used in the drawn picture (dry pen, crayon or watercolor) is left to the availability of the participants, and it will be stated that they prefer colors and drawings that will raise their emotions, focus their drawings and feed positive emotions in the picture to be drawn. After drawing pictures three days before the menstrual cycle and the first day of menstruation (for a total of four days), pain, menstrual symptoms, and perceived stress on the first day of menstruation will be measured using the VAS, MSS, and PSS, respectively.

Control Group: Nursing students with dysmenorrhea in the control group were informed that drawing and listening to music practices would be performed after the initial, second and third month evaluations of the study. In the meantime, it was stated that he should not make any interventions other than her routine applications. At baseline, second, and third month, participants will measure pain, menstrual symptoms, and perceived stress on the first day of the menstrual cycle using the VAS, MSS, and PSS, respectively.

Measures: "Personal Information Form", "Visual Analog Scale (VAS)", "Menstruation Symptom Scale (MSS)" and "Perceived Stress Scale (PSS)" were used in the study.

Personal Information Form: It consists of a total of 36 questions, including socio-demographic characteristics and features related to the menstrual cycle. Within the scope of socio-demographic characteristics; age, height, weight, bki, mother's education level, mother's employment status, father's education level, father's employment status, income status, family type, smoking status, alcohol use status, physical exercise status, place of residence during education life, heavy There are questions such as dominant personality structure, perspective on life. Within the scope of the characteristics related to the menstrual cycle, the first menarche age, the duration of the menstrual cycle, its frequency, the regularity of the menstrual cycle, the reaction of waiting to be menstrual before the menstrual cycle, the feeling of cramp-like pain (dysmenorrhea) in the lower part of the abdomen in the first days of the menstrual cycle, the state of feeling experienced during the menstrual cycle. Problems and coping methods, duration of dysmenorrhea complaint, use of pharmacological treatment method in dysmenorrhea, use of traditional and alternative treatment methods in dysmenorrhea, information source and sharing with a health professional if using, status and frequency of applying to the emergency department with dysmenorrhea complaints are included. The questions were prepared by the researchers in line with the literature, and expert opinion was taken after the questionnaire was prepared.

Visual Analog Scale (VAS): The intensity of menstrual pain will be measured using the VAS, a valid and reliable tool to measure experimental and clinical pain. The VAS is scored on a horizontal line of 10 cm (0=no pain and 10=worst possible pain).

The Menstruation Symptom Scale (MSS): This scale was developed in English by Chesney and Tasto in 1975 to assess menstrual pain and symptoms. It is a widely used scale in the United States and many different countries. The factor structure and usability on adolescents were reassessed and updated. The adaptation of the scale to Turkish was done. Participants are asked to give a number between 1 (never) and 5 (always) for the symptoms they experience about menstruation. The items of the scale are numbered according to the factors set aside for ease of use. 1-13. The items belong to the "Negative effects/somatic complaints" sub-dimension, 14-19. Items included in the "Menstrual pain symptoms" sub-dimension and 20-22. items belong to the sub-dimension "Coping methods". Cronbach's Alpha value is 0.86. It is a five-point Likert-type scale consisting of 22 items. The score obtained from the sub-dimensions is calculated by taking the total score average of the items in the sub-dimensions. The increase in the mean score for the sub-dimensions indicates that the severity of menstrual symptoms related to that sub-dimension increases.

Perceived Stress Scale (PSS): This scale is a self-rating scale developed. The total score that can be obtained from the scale is 32. A high total score from the scale, which consists of 10 items and scored between 0-4, indicates a high level of stress. In this study, the scale whose Turkish validity and reliability study was conducted was used.

Sample size calculation for the primary research question was performed based on a pilot study. Power analysis of this research was done with G*POWER 3.1.9.7 (Power analysis statistical software). In determining the sample size, the value of menstrual pain intensity was taken as the basis. It was determined that 28 individuals from each group would be sufficient to participate in the study, with an effect size of 0.75, margin of error of α=0.05 and minimum power=80% (β=0.2). However, considering the possible missing data, it was decided to include 32 female nursing students in the study by making 10% increase in each group.

ELIGIBILITY:
Inclusion Criteria:

* Has not given birth,
* The ages of 18-25,
* Having a regular menstrual cycle (28±7 days),
* Menstrual pain severity in the previous month is 5 or higher on the Visual Analogue Scale (VAS),
* Having dysmenorrhea,
* Having their written consent,
* Nursing students who volunteered to participate in the study

Exclusion Criteria:

* Hearing loss
* Having chronic disease such as pelvic pathology, neurological, endocrine or psychiatric disease and diabetes mellitus or heart disease,
* Currently using drugs such as antidepressants or oral contraceptives,
* Havingmenstrual irregularity,
* Having mental problems that prevent evaluation and cooperation,
* Obesity, malignant condition, pelvic surgery, pregnancy,
* Using analgesics,
* Using medication or non-drug practices (reiki, meditation, reflexology, acupressure, etc.),
* Nursing students who did not volunteer to participate in the study

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 96 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Pain evaluated using the Visual Analog Scale. | change from before implamentation patent and after 2. and 3. month of practice.
  The intensity of pain is measured using the VAS, a valid and reliable tool for measuring experimental and clinical pain. The VAS is scored on a horizontal line of 10 cm (0=no pain and 10=worst possible pain).
Mensruation symptom evaluated using the Menstruation Symptom Scale (MSS). | change from before implamentation patent and after 2. and 3. month of practice.
  This scale was developed in English by Chesney and Tasto in 1975 to assess menstrual pain and symptoms. It is a widely used scale in the United States and many different countries. In 2009, Negriff et al. The factor structure and usability on adolescents were reassessed and updated. The adaptation of the scale to Turkish was done by Güvenç et al. in 2014. Participants are asked to give a number between 1 (never) and 5 (always) for the symptoms they experience about menstruation. Cronbach's Alpha value is 0.86. It is a five-point Likert-type scale consisting of 22 items. The score obtained from the sub-dimensions is calculated by taking the total score average of the items in the sub-dimensions. The increase in the mean score for the sub-dimensions indicates that the severity of menstrual symptoms related to that sub-dimension increases.
Perceive stress evaluated using the Perceived Stress Scale (PSS). | change from before implamentation patent and after 2. and 3. month of practice.
  This scale is a self-rating scale developed by Cohen, Kamarck, and Mermelstein (1983). The total score that can be obtained from the scale is 32. A high total score from the scale, which consists of 10 items and scored between 0-4, indicates a high level of stress. In this study, the scale whose Turkish validity and reliability study was conducted by Bilge, Öğce, Genç, and Oran (2009) was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kucukkaya B, Basgol S. The effect of listening to music and drawing on coping with dysmenorrhea complaints in nursing students: randomized controlled trial. BMC Womens Health. 2024 Oct 25;24(1):571. doi: 10.1186/s12905-024-03398-0. PMID 39455971